CLINICAL TRIAL: NCT01327651
Title: The ADAPT Study: A Phase II, Randomized, Open-Label, Pharmacokinetic and Behavioral Study of the Use of Intermittent Oral Emtricitabine/Tenofovir Disoproxil Fumarate Pre-Exposure Prophylaxis (PrEP) Pre-Exposure Prophylaxis (PrEP)
Brief Title: The ADAPT Study: Use of Emtricitabine and Tenofovir Disoproxil Fumarate for Pre-Exposure Prophylaxis (PrEP)
Acronym: ADAPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 067 (ADAPT); 10852 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2010-12-01; First posted 2011-04-01 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: Drug Administration Schedule; Nucleoside Reverse Transcriptase Inhibitors; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

STUDY DESIGN:
Intervention Model Description: One arm is daily TDF/FTC. One arm is twice weekly TDF/FTC with a post-exposure dose. One arm is as needed TDF/FTC with a post-exposure dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Daily dosing (Active Comparator): Participants will receive oral FTC/TDF daily.
  Interventions: Drug: Daily dosing
- Time-driven dosing (Experimental): Participants will receive oral FTC/TDF twice weekly with a post-exposure dose.
  Interventions: Drug: Time-driven dosing
- Event-driven dosing (Experimental): Participants will receive oral FTC/TDF before and after a potential exposure to HIV infection.
  Interventions: Drug: Event-driven dosing

INTERVENTIONS:
Drug: Daily dosing — A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate.
  Other Names: Daily; TDF/FTC
  Arms: Daily dosing
Drug: Time-driven dosing — TDF/FTC twice weekly with a post-exposure dose
  Other Names: A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate.
  Arms: Time-driven dosing
Drug: Event-driven dosing — TDF/FTC as needed with a post exposure dose
  Other Names: A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate.
  Arms: Event-driven dosing

SUMMARY:
Pre-exposure prophylaxis (PrEP) is a method of preventing HIV infection through the use of antiretroviral (ARV) medications before exposure to HIV. This study will examine the feasibility of different methods of dosing for a PrEP regimen. Three methods of delivery will be compared: daily, time-based, and event-based.

DETAILED DESCRIPTION:
No single strategy for the prevention of HIV has emerged as consistently used and successful, so multiple strategies have been developed. PrEP involves delivering ARV medications to people before they are exposed to HIV, in order to prevent infection. The optimal method of delivering PrEP has not yet been determined. This study will examine the feasibility of delivering PrEP in three methods. Daily dosing involves receiving ARV medications every day; time-driven dosing involves receiving ARV medications twice weekly plus a post-exposure dose; and event-driven dosing involves receiving ARV medications before and after a potential exposure to HIV. The ARV medication that will be used in this study is a combination pill that contains emtricitabine and tenofovir disoproxil fumarate (FTC/TDF). Recent research studies have shown that, if taken consistently, a daily oral dose of FTC/TDF can reduce the risk of HIV infection.

This study will enroll HIV-uninfected men who have sex with men and transgender women (MSM/TGW) and women who have sex with men (WSM). Participation will last 34 weeks. All participants will be given a combination pill that contains FTC/TDF. For the first 5 weeks, all participants will come to the study clinic weekly to receive a single dose of FTC/TDF.

At Week 6, participants will be randomly assigned to one of three groups. In the daily dosing group, participants will take FTC/TDF once a day. In the time-dosing group, participants will take FTC/TDF twice per week and another dose after sexual intercourse (a post-exposure dose). In the event-dosing group, participants will take FTC/TDF before and after sexual intercourse. During this part of the study, participants will be given FTC/TDF to take on their own. Every week, from Week 6 to Week 29, study officials will call to ask questions about how many pills participants have taken and when they have had sexual intercourse. Participants will also complete computer-assisted self-interviews (CASIs).

Study visits will occur at enrollment, once a week for the first 5 weeks, and then once a month until Week 34. Assessment will include recording of medical history, completing an interview about sexual practices and background, and collection of blood, urine, and hair samples. Select study visits will include vaginal practices assessment (including use of lubricants and vaginal cleansing practices), family planning assessments (for women), and sex hormones assessments (for men).

Participants who acquire HIV infection during the study will discontinue study product. These participants will continue to be followed after enrollment at Weeks 4, 6, 10, 14, 18, 22, 26, 30, and every 12 weeks thereafter, as appropriate, until the last study participant completes follow-up at the study site. Participants whose first reactive HIV rapid test is at Week 34 who are later confirmed to be HIV infected will also be followed every 12 weeks after their Week 30 visit until the last study participant completes follow-up at the study site. Participants who acquire HIV infection during the study will undergo select protocol procedures and will receive counseling and referrals for HIV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Literacy in one of the study languages (Thai, Xhosa, and/or English)
* Able to provide written informed consent
* Able to provide weekly telephonic updates
* Within 70 days of enrollment:

  1. Serum creatinine less than or equal to the upper limit of normal (ULN) and calculated creatinine clearance of at least 70 mL/min by the Cockcroft-Gault formula. More information on this criterion can be found in the protocol.
  2. Serum phosphate greater than or equal to the lower limit of normal (LLN)
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 2 times ULN
  4. Hemoglobin greater than 10 g/dL
  5. Hepatitis B surface antigen (HBsAg)-negative
  6. Willing and able to provide adequate locator information

Inclusion Criteria for MSM/TGW:

* Male at birth
* Reporting anal intercourse and/or receptive neovaginal intercourse with at least one man or transgender woman in the past 6 months
* One or more of the following risk factors for HIV acquisition in the past 6 months according to self-report: sexual intercourse with more than one man or transgender woman; history of an acute sexually transmitted infection (STI); sex in exchange for money, goods, or favors; condomless intercourse (oral, anal, vaginal, or neovaginal) with a partner known to be HIV-infected or of unknown HIV infection status according to self report

Inclusion Criteria for Women Who Have Sex With Men (WSM):

* Female at birth or self identify as female
* Not pregnant or breastfeeding
* Not able to or not intending to become pregnant during the next year
* If able to become pregnant, self reported use of an effective method of contraception at Enrollment, and intending to use an effective method for the next 34 weeks
* One or more of the following risk factors for HIV acquisition in the past 6 months according to self report: sexual intercourse with more than one man; history of an acute STI; sex in exchange for money, goods or favors; condomless intercourse (oral, anal, or vaginal) with a partner known to be HIV-infected or of unknown HIV infection status

Exclusion Criteria:

* Proteinuria 2+ or greater at screening
* Glucosuria 2+ or greater at screening
* Serious and active medical or mental illness
* One or both HIV rapid tests is reactive at screening or enrollment, regardless of subsequent HIV diagnostic test results
* Signs or symptoms suggestive of acute HIV infection
* Use of hypoglycemic agents for diabetes or agents with known nephrotoxic potential
* Use of ARV therapy (e.g., for post-exposure prophylaxis [PEP] or PrEP) in the 90 days prior to study entry
* Serum phosphate level below site laboratory LLN
* Current participation (or participation within 3 months of screening) in any HIV prevention study
* Previous or current participation in the active arm of an HIV vaccine trial
* Acute or chronic hepatitis B (HBV) infection (refers to chronic active HBV infection evidenced by a positive test for hepatitis B surface antigen (HBsAg)
* Presence of a psychological or social condition or an addictive disorder that would preclude compliance with the protocol
* Any other reason or condition that in the opinion of the investigator would interfere with participation, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Grant, MD, MPH, Study Chair — University of California, San Francisco; Frits van Griensven, PhD, MPH, Study Chair — School of Medicine, University of California at San Francisco
Locations (3):
- Harlem Prevention Center CRS, New York, New York, United States
- Emavundleni CRS, Cape Town, Western Cape, South Africa
- Silom Community Clinic CRS, Nonthaburi, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Derived] Hughes JP, Williamson BD, Krakauer C, Chau G, Ortiz B, Wakefield J, Hendrix C, Amico KR, Holtz TH, Bekker LG, Grant R. Combining information to estimate adherence in studies of pre-exposure prophylaxis for HIV prevention: Application to HPTN 067. Stat Med. 2022 Mar 15;41(6):1120-1136. doi: 10.1002/sim.9321. Epub 2022 Jan 25. PMID 35080038
- [Derived] Holtz TH, Chitwarakorn A, Hughes JP, Curlin ME, Varangrat A, Li M, Amico KR, Mock PA, Grant RM; Thai HPTN 067/ADAPT Study Team. HPTN 067/ADAPT: Correlates of Sex-Related Pre-exposure Prophylaxis Adherence, Thai Men Who Have Sex With Men, and Transgender Women, 2012-2013. J Acquir Immune Defic Syndr. 2019 Oct 1;82(2):e18-e26. doi: 10.1097/QAI.0000000000002131. PMID 31490342
- [Derived] Grant RM, Mannheimer S, Hughes JP, Hirsch-Moverman Y, Loquere A, Chitwarakorn A, Curlin ME, Li M, Amico KR, Hendrix CW, Anderson PL, Dye BJ, Marzinke MA, Piwowar-Manning E, McKinstry L, Elharrar V, Stirratt M, Rooney JF, Eshleman SH, McNicholl JM, van Griensven F, Holtz TH. Daily and Nondaily Oral Preexposure Prophylaxis in Men and Transgender Women Who Have Sex With Men: The Human Immunodeficiency Virus Prevention Trials Network 067/ADAPT Study. Clin Infect Dis. 2018 May 17;66(11):1712-1721. doi: 10.1093/cid/cix1086. PMID 29420695
- [Derived] Bekker LG, Roux S, Sebastien E, Yola N, Amico KR, Hughes JP, Marzinke MA, Hendrix CW, Anderson PL, Elharrar V, Stirratt M, Rooney JF, Piwowar-Manning E, Eshleman SH, McKinstry L, Li M, Dye BJ, Grant RM; HPTN 067 (ADAPT) study team. Daily and non-daily pre-exposure prophylaxis in African women (HPTN 067/ADAPT Cape Town Trial): a randomised, open-label, phase 2 trial. Lancet HIV. 2018 Feb;5(2):e68-e78. doi: 10.1016/S2352-3018(17)30156-X. Epub 2017 Oct 3. PMID 28986029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled men, and transgender women, who have sex with men at a community clinic and clinical research site (CRS) in Bangkok, Thailand, and a CRS in Harlem in New York City, USA. Women were enrolled at a study site in Cape Town, South Africa. The last participant was enrolled in May of 2014
Pre-assignment Details: Of the 902 screened participants, 622 were eligible to be enrolled into the study, and participated in a 6-week lead-in period of directly observed dosing (DOD) of one tablet once-weekly of FTC/TDF for five observed doses followed by 1-week off drug. 86% (N=536) completed the lead-in period and were randomized to the three arms.
Groups:
- Daily Dosing, Cape Town: Cape Town participants will receive oral FTC/TDF daily. Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors.
- Time-driven Dosing, Cape Town: Cape Town participants will receive oral FTC/TDF twice weekly with a post-exposure dose.
  Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors.
- Event-driven Dosing, Cape Town: Cape Town participants will receive oral FTC/TDF before and after a potential exposure to HIV infection.
  Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors.
- Daily Dosing, Bangkok: Bangkok participants will receive oral FTC/TDF daily. Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors.
- Time-driven Dosing, Bangkok: Bangkok participants will receive oral FTC/TDF twice weekly with a post-exposure dose.
  Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors
- Event-driven Dosing, Bangkok: Bangkok participants will receive oral FTC/TDF before and after a potential exposure to HIV infection.
  Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors.
- Daily Dosing, Harlem: Harlem participants will receive oral FTC/TDF daily. Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors.
- Time-driven Dosing, Harlem: Harlem participants will receive oral FTC/TDF twice weekly with a post-exposure dose.
  Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors.
- Event-driven Dosing, Harlem: Harlem participants will receive oral FTC/TDF before and after a potential exposure to HIV infection.
  Emtricitabine/Tenofovir Disoproxil Fumarate (FTC/TDF): A fixed-dose combination of emtricitabine and tenofovir disoproxil fumarate, two nucleoside reverse transcriptase inhibitors.
Period: Self-administered Dosing Period
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Started (Week 6 (Randomization visit)) | 60 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
Week 10 | 59 | 58 | 60 | 60 | 59 | 59 | 57 | 57 | 56
Week 14 | 59 | 55 | 57 | 60 | 58 | 59 | 54 | 51 | 54
Week 18 | 57 | 56 | 56 | 60 | 57 | 59 | 53 | 49 | 53
Week 22 | 59 | 56 | 55 | 58 | 56 | 59 | 50 | 50 | 51
Week 26 | 58 | 56 | 53 | 57 | 56 | 58 | 50 | 51 | 49
Completed (Week 30) | 56 | 56 | 56 | 57 | 56 | 59 | 49 | 50 | 49
Not Completed | 4 | 3 | 4 | 3 | 3 | 0 | 10 | 10 | 11
Not completed — Lost to Follow-up | 3 | 2 | 4 | 2 | 3 | 0 | 8 | 9 | 10
Not completed — Ineligible (retrospective result) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 1
Period: Post Study Follow-up
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Started (Week 30) | 56 | 56 | 56 | 57 | 56 | 59 | 49 | 50 | 49
Completed (Week 34) | 56 | 55 | 55 | 57 | 56 | 59 | 45 | 49 | 47
Not Completed | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Population: For daily dosing arm in Cape Town, we dropped one participant from analysis, since retrospective test of HIV infection in central lab shows that this participant was seroconverted on week 6(randomization week), so she was not eligible to be randomized. Because of this, total baseline population dropped from 536 to 535.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem | Total
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60 | 535
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25 [21 to 37] | 26 [21 to 33] | 25 [21 to 37] | 31 [28 to 34] | 28 [25 to 35] | 31 [27 to 34] | 28 [23 to 43] | 31 [24 to 41] | 32 [24 to 46] | 29 [24 to 37]
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 26 | 24 | 26 | 8 | 12 | 8 | 19 | 17 | 17 | 157
  25-29 years | 14 | 15 | 8 | 13 | 19 | 16 | 13 | 11 | 8 | 117
  30-39 years | 10 | 11 | 16 | 36 | 23 | 28 | 11 | 12 | 14 | 161
  40+ years | 9 | 9 | 10 | 3 | 5 | 7 | 16 | 20 | 21 | 100
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 59 | 59 | 60 | 0 | 0 | 0 | 0 | 0 | 0 | 178
  Male | 0 | 0 | 0 | 59 | 58 | 59 | 57 | 59 | 58 | 350
  Transgender woman | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 5
  Gender queer | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  Less than secondary | 38 | 39 | 39 | 0 | 1 | 1 | 16 | 18 | 7 | 159
  Secondary and above | 21 | 20 | 21 | 60 | 58 | 58 | 43 | 42 | 53 | 376
Number of sex partners in the past 3 months [Median (Inter-Quartile Range); unit: sex partners] — Median number of sex partners in the past 3 months, measured at baseline
  sex partners | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 3 [2 to 10] | 3 [1 to 10] | 3 [2 to 5] | 3 [2 to 5] | 3 [2 to 6] | 4 [2 to 7] | 2 [1 to 5]
Number of anal intercourse without a condom [Median (Inter-Quartile Range); unit: anal intercourse] | 2 [0 to 7] | 2 [0 to 5] | 1 [0 to 4] | 0 [0 to 5] | 0 [0 to 3] | 0 [0 to 0] | 3 [0 to 5] | 3 [1 to 10] | 5 [1 to 9] | 1 [0 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Sexual Exposures Covered by Pre- and Post-exposure Dosing
Description: Coverage will be determined based on the adjusted electronic and self-reported pill-use data. Specifically, a sex act will be considered as "covered" if at least one pill is taken 96 hours prior the sexual activity and at least one additional pill is taken within 24 hours after the sexual activity. If participant only took pill before the sexual activity (within 96 hours), but no pill taken after sexual activity (within 24 hours), then we considered it as pre-exposure covered. likewise, if participant only took pill after sexual activity (within 24 hours), but did not taken pill before sexual activity (within 96 hours), then we considered it as post-exposure covered. If participant did not taken pill before and after sexual activity, then it was considered as not covered. Note that the same pill can be both pre-exposure dose and a post-exposure dose if events are closely spaced. At no time should a participant in the intermittent arm be taking more pills than the daily arm.
Time Frame: From week 6 (randomization week) to week 30 (end of self-administered dosing)
Population: For Cape Town daily dosing arm, there are originally 60 participants, but 1 participant was later found to be HIV infected on or before randomization visit, which should make this participant not eligible for the study analysis, so we removed this participant from this table. Given this, we left 59 participants in Cape Town daily dosing arm
Measure: Number; unit: percentage of sexual exposures
Units Other Than Participants: sexual exposures
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
Number analyzed (sexual exposures) | 1952 | 1074 | 1542 | 1485 | 1337 | 1018 | 1081 | 1311 | 1502
percentage of sexual exposures
  % completely covered | 75 | 56 | 52 | 85 | 84 | 74 | 66 | 47 | 52
  % pre-exposure coverage | 21 | 30 | 33 | 11 | 12 | 19 | 24 | 30 | 29
  % post-exposure coverage | 1 | 9 | 8 | 1 | 3 | 5 | 2 | 8 | 6
  % uncovered | 3 | 5 | 7 | 3 | 1 | 3 | 8 | 15 | 13

2. Primary Outcome: The (Minimum) Total Number of Pills Needed for 100% Coverage Over the Follow-up Period (Based on Randomization Arm and Self-reported Sexual History in the Weekly Interviews)
Description: Below I reported the number of sex acts as reported based on the adjusted electronic and self-reported sexual activity data, also the number of pills needed for 100% coverage. 100% coverage means all sex events (excluding oral sex) are "covered"; Note: sex act is considered as "covered" if at least one pill is taken 96 hours prior the sexual activity and at least one additional pill is taken within 24 hours after the sexual activity (same coverage definition for all three arms)
Time Frame: From week 6 (randomization week) to week 30 (end of self-administered dosing)
Population: as for outcome 1
Measure: Number; unit: Number of pills needed for 100% coverage
Units Other Than Participants: sexual exposure
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
Number analyzed (sexual exposure) | 1952 | 1074 | 1542 | 1485 | 1337 | 1018 | 1081 | 1311 | 1502
Number of pills needed for 100% coverage | 2097 | 1552 | 1906 | 1746 | 1573 | 1268 | 1244 | 1390 | 1582

3. Primary Outcome: The Total Pills Actually Used Over the Follow-up Period
Description: The total pills actually used over the follow-up period was calculated based on the adjusted electronic and self-reported pill-use data. It could be more or less than required by study design
Time Frame: From week 6 (randomization week) to week 30 (end of self-administered dosing)
Population: as for outcome 1
Measure: Number; unit: Number of pills actually used
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
Number of pills actually used | 7349 | 2852 | 2000 | 8285 | 3713 | 2157 | 5507 | 2468 | 2356

4. Primary Outcome: Self-reported Side Effect or Symptom Scores
Description: The self-reported symptom/side effect scores for common symptoms/side effects including headache, dizziness, cramping, abdominal pain, and flatulence. Collected during clinic visits. All the presented numbers are the percent of visits with each side effects
Time Frame: From week 6 (randomization week) to week 30 (end of self-administered dosing)
Population: as for outcome 1
Measure: Number; unit: percent of visits between week 6 to 30
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
percent of visits between week 6 to 30
  Neurologic side effect | 12.4 | 6.0 | 7.8 | 14.2 | 14.3 | 13.3 | 6.1 | 3.3 | 4.5
  Gastrointestinal side effects | 10.6 | 8.8 | 5.4 | 13.1 | 8.5 | 10.5 | 8 | 5.8 | 7.1

5. Secondary Outcome: Measurement of TFV-DP (Tenofovir Diphosphate) in PBMC (Peripheral Blood Mononuclear Cell)
Description: Below we presented the percentages of total cohort with TFV-DP concentrations consistent with >=2 pills/week in women who also report sex in the last 7 day for each arm. For Cape Town and Bangkok, TFV-DP in PBMC was analyzed, for Harlem site, the TFV-DP in DBS (dried blood spot) was analyzed. Note: PBMC >5.2 fmol/10^6 cells is considered as participants taken >=2 tablets per week; DBS >=326 fmol/punch is considered as participants taken >=2 tablets per week
Time Frame: week 10, 18 and 30, which is 4 weeks, 12 weeks, and 24 weeks after randomization
Population: Note: Not all participants were available to be analyzed at each visits below, this could be due to missed visit, drug concentration was missing, or participants did not report to have any sex in the last 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
Participants
  Week 10: number analyzed (Participants) | 40 | 23 | 37 | 31 | 29 | 30 | 23 | 23 | 27
  Week 10 | 33 | 16 | 25 | 31 | 29 | 30 | 13 | 8 | 5
  Week 18: number analyzed (Participants) | 39 | 25 | 30 | 29 | 30 | 26 | 27 | 27 | 21
  Week 18 | 29 | 16 | 10 | 28 | 30 | 24 | 11 | 10 | 3
  Week 30: number analyzed (Participants) | 29 | 24 | 31 | 23 | 19 | 14 | 18 | 18 | 18
  Week 30 | 19 | 13 | 12 | 22 | 18 | 13 | 9 | 3 | 3

6. Secondary Outcome: A Listing of Adverse Events (AEs) by Grade, Relationship to Study Product, and Arm
Description: Only the listing of adverse events (AEs) by grade and arm are presented here. See outcome measure 10 for the listing of AE by relationship to study product
Time Frame: From week 6 (randomization week) to week 30 (end of self-administered dosing)
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
Participants
  Blood and lymphatic system disorders : Mild: Mild | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Blood and lymphatic system disorders : Mild: Moderate | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Blood and lymphatic system disorders : Mild: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood and lymphatic system disorders : Mild: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood and lymphatic system disorders : Mild: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood and lymphatic system disorders : Mild: None | 57 | 57 | 59 | 60 | 59 | 59 | 57 | 58 | 58
  Cardiac disorders: Mild | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0
  Cardiac disorders: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cardiac disorders: None | 59 | 59 | 59 | 58 | 58 | 58 | 58 | 60 | 60
  Ear and labyrinth disorders: Mild | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Ear and labyrinth disorders: Moderate | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Ear and labyrinth disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ear and labyrinth disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ear and labyrinth disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ear and labyrinth disorders: None | 58 | 56 | 60 | 59 | 59 | 58 | 58 | 60 | 59
  Eye disorders: Mild | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 2
  Eye disorders: Moderate | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders: None | 55 | 57 | 59 | 59 | 59 | 59 | 57 | 60 | 58
  Gastrointestinal disorders: Mild | 18 | 17 | 18 | 24 | 22 | 23 | 28 | 27 | 28
  Gastrointestinal disorders: Moderate | 8 | 9 | 10 | 6 | 1 | 3 | 1 | 2 | 1
  Gastrointestinal disorders: Severe | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Gastrointestinal disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders: None | 33 | 32 | 32 | 30 | 35 | 32 | 30 | 31 | 31
  General disorders and administration site conditio: Mild | 9 | 5 | 7 | 10 | 16 | 11 | 10 | 10 | 8
  General disorders and administration site conditio: Moderate | 0 | 2 | 5 | 0 | 0 | 1 | 2 | 1 | 0
  General disorders and administration site conditio: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  General disorders and administration site conditio: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  General disorders and administration site conditio: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  General disorders and administration site conditio: None | 50 | 52 | 48 | 50 | 43 | 47 | 46 | 49 | 52
  Hepatobiliary disorders: Mild | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hepatobiliary disorders: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hepatobiliary disorders: Severe | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hepatobiliary disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hepatobiliary disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hepatobiliary disorders: None | 59 | 58 | 60 | 60 | 58 | 59 | 59 | 60 | 60
  Immune system disorders: Mild | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Immune system disorders: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Immune system disorders: Severe | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Immune system disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Immune system disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Immune system disorders: None | 59 | 59 | 58 | 60 | 59 | 59 | 59 | 59 | 59
  Infections and infestations: Mild | 11 | 10 | 15 | 22 | 33 | 28 | 22 | 21 | 21
  Infections and infestations: Moderate | 25 | 25 | 21 | 8 | 6 | 10 | 0 | 0 | 1
  Infections and infestations: Severe | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 1
  Infections and infestations: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations: None | 23 | 24 | 24 | 27 | 19 | 19 | 37 | 39 | 37
  Injury, poisoning and procedural complications: Mild | 7 | 5 | 11 | 16 | 15 | 14 | 17 | 18 | 14
  Injury, poisoning and procedural complications: Moderate | 3 | 2 | 1 | 0 | 2 | 1 | 2 | 1 | 0
  Injury, poisoning and procedural complications: Severe | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 1
  Injury, poisoning and procedural complications: Potentically Life Threatening | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Injury, poisoning and procedural complications: None | 48 | 51 | 46 | 44 | 41 | 44 | 38 | 41 | 45
  Investigations: Mild | 13 | 15 | 13 | 18 | 9 | 7 | 8 | 6 | 6
  Investigations: Moderate | 5 | 6 | 3 | 5 | 2 | 3 | 1 | 2 | 2
  Investigations: Severe | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 0
  Investigations: Potentically Life Threatening | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Investigations: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Investigations: None | 41 | 38 | 43 | 35 | 47 | 48 | 50 | 50 | 52
  Metabolism and nutrition disorders: Mild | 0 | 3 | 7 | 0 | 1 | 0 | 3 | 4 | 5
  Metabolism and nutrition disorders: Moderate | 6 | 5 | 10 | 0 | 0 | 1 | 2 | 3 | 4
  Metabolism and nutrition disorders: Severe | 3 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Metabolism and nutrition disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Metabolism and nutrition disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Metabolism and nutrition disorders: None | 50 | 49 | 43 | 60 | 58 | 58 | 52 | 53 | 51
  Musculoskeletal and connective tissue disorders: Mild | 6 | 6 | 9 | 13 | 15 | 13 | 13 | 11 | 9
  Musculoskeletal and connective tissue disorders: Moderate | 3 | 2 | 1 | 4 | 1 | 2 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Musculoskeletal and connective tissue disorders: None | 50 | 51 | 50 | 43 | 43 | 44 | 46 | 49 | 51
  Nervous system disorders: Mild | 17 | 14 | 19 | 17 | 18 | 22 | 16 | 10 | 17
  Nervous system disorders: Moderate | 15 | 11 | 12 | 3 | 0 | 1 | 1 | 2 | 0
  Nervous system disorders: Severe | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Nervous system disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders: None | 27 | 34 | 29 | 39 | 41 | 36 | 42 | 47 | 43
  Pregnancy, puerperium and perinatal conditions: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pregnancy, puerperium and perinatal conditions: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pregnancy, puerperium and perinatal conditions: Severe | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pregnancy, puerperium and perinatal conditions: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pregnancy, puerperium and perinatal conditions: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pregnancy, puerperium and perinatal conditions: None | 58 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
  Psychiatric disorders: Mild | 1 | 3 | 2 | 8 | 10 | 8 | 10 | 9 | 7
  Psychiatric disorders: Moderate | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
  Psychiatric disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Psychiatric disorders: Potentically Life Threatening | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  Psychiatric disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Psychiatric disorders: None | 55 | 56 | 56 | 52 | 49 | 51 | 46 | 48 | 52
  Renal and urinary disorders: Mild | 10 | 11 | 11 | 1 | 3 | 2 | 12 | 6 | 7
  Renal and urinary disorders: Moderate | 4 | 2 | 3 | 0 | 1 | 1 | 0 | 4 | 1
  Renal and urinary disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Renal and urinary disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Renal and urinary disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Renal and urinary disorders: None | 45 | 46 | 46 | 59 | 55 | 56 | 47 | 50 | 52
  Reproductive system and breast disorders: Mild | 13 | 17 | 17 | 0 | 0 | 1 | 1 | 2 | 3
  Reproductive system and breast disorders: Moderate | 7 | 8 | 8 | 0 | 0 | 1 | 0 | 0 | 0
  Reproductive system and breast disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reproductive system and breast disorders: Potentically Life Threatening | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Reproductive system and breast disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Reproductive system and breast disorders: None | 39 | 34 | 34 | 60 | 59 | 57 | 58 | 58 | 57
  Respiratory, thoracic and mediastinal disorders: Mild | 5 | 5 | 9 | 36 | 23 | 29 | 18 | 19 | 18
  Respiratory, thoracic and mediastinal disorders: Moderate | 5 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders: None | 49 | 52 | 50 | 24 | 36 | 29 | 41 | 41 | 42
  Skin and subcutaneous tissue disorders: Mild | 6 | 8 | 8 | 8 | 15 | 10 | 8 | 5 | 5
  Skin and subcutaneous tissue disorders: Moderate | 3 | 3 | 4 | 2 | 0 | 3 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders: Severe | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders: None | 49 | 48 | 48 | 50 | 44 | 46 | 51 | 55 | 55
  Social circumstances: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Social circumstances: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Social circumstances: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Social circumstances: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Social circumstances: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Social circumstances: None | 58 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
  Vascular disorders: Mild | 2 | 3 | 1 | 0 | 0 | 1 | 2 | 0 | 0
  Vascular disorders: Moderate | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vascular disorders: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vascular disorders: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vascular disorders: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vascular disorders: None | 56 | 55 | 59 | 60 | 59 | 58 | 57 | 60 | 60
  Neoplasms benign, malignant, and unspecified: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neoplasms benign, malignant, and unspecified: Moderate | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Neoplasms benign, malignant, and unspecified: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neoplasms benign, malignant, and unspecified: Potentically Life Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neoplasms benign, malignant, and unspecified: Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neoplasms benign, malignant, and unspecified: None | 59 | 59 | 60 | 60 | 59 | 58 | 59 | 60 | 60

7. Secondary Outcome: A Listing, by Arm, of Drug Resistance Test Results and Plasma HIV RNA Levels Among All Participants Who Seroconvert While on Study
Description: Only the cross table between drug resistance by arm are presented here. See outcome measure 11 for the listing of plasma HIV RNA levels, and outcome measure 12 for the listing of drug resistance test by arm among all participants who seroconvert while on study.
Time Frame: From enrollment to week 30 (end of self-administered dosing)
Population: Data is collected for plasma HIV RNA levels among all participants who seroconvert while on study, but this secondary analysis has not been carried out yet, so no outcome measure is presented here
Measure: Count of Participants; unit: Participants
Groups:
- Cape Town, South Africa: The University of Cape Town in Cape Town is the IRB of record for the Cape Town site
- Bangkok, Thailand: The Institutional Review Board, Human Research Protection Office, US Centers for Disease Control and Prevention and the Ethical Review Committee for Research in Human Subjects, Department of Medical Sciences, Ministry of Public Health, Thailand are the IRBs of record for the Bangkok site
- Harlem, United States: Columbia University Medical Center Institutional Review Board in New York is the IRB of record for the New York site.
Arm/Group | Cape Town, South Africa | Bangkok, Thailand | Harlem, United States
Number analyzed (Participants) | 191 | 193 | 238
Participants
  Before Randomization: Drug Resistance | 1 | 0 | 1
  Before Randomization: No Drug Resistance | 190 | 193 | 237
  After Randomization (Daily dosing): number analyzed (Participants) | 59 | 60 | 59
  After Randomization (Daily dosing): Drug Resistance | 0 | 0 | 0
  After Randomization (Daily dosing): No Drug Resistance | 59 | 60 | 59
  After Randomization (Time-driven dosing): number analyzed (Participants) | 59 | 59 | 60
  After Randomization (Time-driven dosing): Drug Resistance | 1 | 0 | 0
  After Randomization (Time-driven dosing): No Drug Resistance | 58 | 59 | 60
  After Randomization (Event-driven dosing): number analyzed (Participants) | 60 | 59 | 60
  After Randomization (Event-driven dosing): Drug Resistance | 0 | 0 | 0
  After Randomization (Event-driven dosing): No Drug Resistance | 60 | 59 | 60

8. Secondary Outcome: The Percentage of Correctly Timed Adherence (Number of Pills Taken Within the Recommended Time Frame/Number of Pills Recommended) During 24 Weeks of Follow-up Based on Weekly Interviews and Adjusted EDM (Electronic Drug Monitoring) Data
Time Frame: From week 6 (randomization week) to week 30 (end of self-administered dosing)
Population: as for outcome 1
Measure: Number; unit: % of Correctly Timed Adherence
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
% of Correctly Timed Adherence | 75 | 65 | 53 | 85 | 79 | 65 | 65 | 47 | 41

9. Secondary Outcome: The Proportion of Participants Who Discontinue All PrEP Use Based on Self-report Via CASI or Weekly Interviews
Time Frame: From Week 6 to Week 30
Population: Number of participants had product hold or product discontinuation log
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 7 | 7 | 8 | 12 | 3 | 5 | 2 | 7 | 2
Participants
  Pregnancy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  HIV-positive result | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  Other adverse experience | 6 | 3 | 5 | 6 | 2 | 1 | 1 | 3 | 0
  Other | 1 | 2 | 1 | 5 | 1 | 4 | 0 | 4 | 2

10. Secondary Outcome: A Listing of Adverse Events (AEs) by Grade, Relationship to Study Product, and Arm
Description: Only the listing of AE related to study product are presented here. See outcome measure 6 for the listing of adverse events (AEs) by grade and arm.
Time Frame: From week 6 (randomization week) to week 30 (end of self-administered dosing)
Population: Below "Number analyzed" population only included the participants who had below adverse events, and the number next to it represent the number of participants had the corresponding AE that was related to the study product
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Number analyzed (Participants) | 59 | 59 | 60 | 60 | 59 | 59 | 59 | 60 | 60
Participants
  Blood and lymphatic system disorders: number analyzed (Participants) | 2 | 2 | 1 | 0 | 0 | 0 | 2 | 2 | 2
  Blood and lymphatic system disorders | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Cardiac disorders: number analyzed (Participants) | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0
  Cardiac disorders | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Ear and labyrinth disorders: number analyzed (Participants) | 1 | 3 | 0 | 1 | 0 | 1 | 1 | 0 | 1
  Ear and labyrinth disorders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders: number analyzed (Participants) | 4 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 2
  Eye disorders | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders: number analyzed (Participants) | 26 | 27 | 28 | 30 | 24 | 27 | 29 | 29 | 29
  Gastrointestinal disorders | 18 | 17 | 24 | 9 | 1 | 2 | 13 | 13 | 16
  General disorders and administration site conditio: number analyzed (Participants) | 9 | 7 | 12 | 10 | 16 | 12 | 13 | 11 | 8
  General disorders and administration site conditio | 4 | 1 | 6 | 1 | 1 | 0 | 3 | 9 | 4
  Hepatobiliary disorders: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hepatobiliary disorders | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Immune system disorders: number analyzed (Participants) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
  Immune system disorders | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Infections and infestations: number analyzed (Participants) | 36 | 35 | 36 | 33 | 40 | 40 | 22 | 21 | 23
  Infections and infestations | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
  Injury, poisoning and procedural complications: number analyzed (Participants) | 11 | 8 | 14 | 16 | 18 | 15 | 21 | 19 | 15
  Injury, poisoning and procedural complications | 3 | 4 | 7 | 10 | 7 | 10 | 13 | 16 | 10
  Investigations: number analyzed (Participants) | 18 | 21 | 17 | 25 | 12 | 11 | 9 | 10 | 8
  Investigations | 10 | 13 | 12 | 23 | 12 | 10 | 9 | 9 | 7
  Metabolism and nutrition disorders: number analyzed (Participants) | 9 | 10 | 17 | 0 | 1 | 1 | 7 | 7 | 9
  Metabolism and nutrition disorders | 2 | 5 | 6 | 0 | 1 | 1 | 4 | 5 | 5
  Musculoskeletal and connective tissue disorders: number analyzed (Participants) | 9 | 8 | 10 | 17 | 16 | 15 | 13 | 11 | 9
  Musculoskeletal and connective tissue disorders | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3
  Neoplasms benign, malignant, and unspecified: number analyzed (Participants) | 59 | 59 | 60 | 0 | 0 | 1 | 0 | 0 | 0
  Neoplasms benign, malignant, and unspecified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nervous system disorders: number analyzed (Participants) | 32 | 25 | 31 | 21 | 18 | 23 | 17 | 13 | 17
  Nervous system disorders | 17 | 17 | 21 | 3 | 2 | 1 | 7 | 4 | 5
  Pregnancy, puerperium and perinatal conditions: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pregnancy, puerperium and perinatal conditions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Psychiatric disorders: number analyzed (Participants) | 4 | 3 | 4 | 8 | 10 | 8 | 13 | 12 | 8
  Psychiatric disorders | 3 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 3
  Renal and urinary disorders: number analyzed (Participants) | 14 | 13 | 14 | 1 | 4 | 3 | 12 | 10 | 8
  Renal and urinary disorders | 10 | 5 | 10 | 0 | 1 | 2 | 8 | 9 | 4
  Reproductive system and breast disorders: number analyzed (Participants) | 20 | 25 | 26 | 0 | 0 | 2 | 1 | 2 | 3
  Reproductive system and breast disorders | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders: number analyzed (Participants) | 10 | 7 | 10 | 36 | 23 | 30 | 18 | 19 | 18
  Respiratory, thoracic and mediastinal disorders | 2 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0
  Skin and subcutaneous tissue disorders: number analyzed (Participants) | 10 | 11 | 12 | 10 | 15 | 13 | 8 | 5 | 5
  Skin and subcutaneous tissue disorders | 4 | 5 | 3 | 2 | 0 | 2 | 1 | 2 | 0
  Social circumstances: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Social circumstances | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vascular disorders: number analyzed (Participants) | 3 | 4 | 1 | 0 | 0 | 1 | 2 | 0 | 0
  Vascular disorders | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

11. Secondary Outcome: A Listing, by Arm, of Drug Resistance Test Results and Plasma HIV RNA Levels Among All Participants Who Seroconvert While on Study
Description: Only the listing of plasma HIV RNA levels among all participants who seroconvert while on study are presented here. See outcome measure 12 for the listing of drug resistance test by arm.
Time Frame: From Enrollment to week 30 (end of self-administered dosing)
Population: Below, each seroconverted participants' plasma HIV RNA levels at all visits with test results are presented
Measure: Number; unit: viral load
Groups:
- Cape Town, South Africa, Seroconverted Participant #1: #1 seroconverted participants in Cape Town, South Africa, not randomized
- Cape Town, South Africa, Seroconverted Participant #2: #2 seroconverted participants in Cape Town, South Africa, not randomized
- Cape Town, South Africa, Seroconverted Participant #3: #3 seroconverted participants in Cape Town, South Africa, not randomized
- Cape Town, South Africa, Seroconverted Participant #4: #4 seroconverted participants in Cape Town, South Africa, daily arm
- Cape Town, South Africa, Seroconverted Participant #5: #5 seroconverted participants in Cape Town, South Africa, time-driven arm
- Cape Town, South Africa, Seroconverted Participant #6: #6 seroconverted participants in Cape Town, South Africa, time-driven arm
- Cape Town, South Africa, Seroconverted Participant #7: #7 seroconverted participants in Cape Town, South Africa, event-driven arm
- Cape Town, South Africa, Seroconverted Participant #8: #8 seroconverted participants in Cape Town, South Africa, event-driven arm
- Bangkok, Thailand, Seroconverted Participant #1: #1 seroconverted participants in Bangkok, Thailand, not randomized
- Bangkok, Thailand, Seroconverted Participant #2: #2 seroconverted participants in Bangkok, Thailand, not randomized
- Harlem, United States, Seroconverted Participant #1: #1 seroconverted participants in Harlem, United States, not randomized
- Harlem, United States, Seroconverted Participant #2: #2 seroconverted participants in Harlem, United States, daily arm
Arm/Group | Cape Town, South Africa, Seroconverted Participant #1 | Cape Town, South Africa, Seroconverted Participant #2 | Cape Town, South Africa, Seroconverted Participant #3 | Cape Town, South Africa, Seroconverted Participant #4 | Cape Town, South Africa, Seroconverted Participant #5 | Cape Town, South Africa, Seroconverted Participant #6 | Cape Town, South Africa, Seroconverted Participant #7 | Cape Town, South Africa, Seroconverted Participant #8 | Bangkok, Thailand, Seroconverted Participant #1 | Bangkok, Thailand, Seroconverted Participant #2 | Harlem, United States, Seroconverted Participant #1 | Harlem, United States, Seroconverted Participant #2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
viral load
  Enrollment: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Enrollment | 20 |  |  |  |  |  |  |  |  |  |  |
  Day 3: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Day 3 | 400 | 400 |  |  |  |  |  |  | 40 | 78450 | 400 |
  Week 4: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Week 4 | 3460 | 3667690 |  |  |  |  |  |  | 749590 | 710 | 40900 |
  Week 5: number analyzed (Participants) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Week 5 | 5732050 | 3938670 |  |  |  |  |  |  |  | 1570 |  |
  Week 6: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Week 6 |  |  |  | 400 |  |  |  |  | 92960 | 5070 | 83260 |
  Week 10: number analyzed (Participants) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Week 10 | 416070 | 93040 |  | 400 |  |  |  |  | 1799950 |  |  |
  Week 14: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
  Week 14 |  | 93660 |  | 400 |  | 2100 |  |  | 119720 |  |  | 1567040
  Week 18: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
  Week 18 |  | 114520 |  | 650 |  | 3710 | 83010 |  | 127330 |  |  | 73030
  Week 22: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Week 22 |  | 178210 |  | 400 | 5887760 | 127480 | 136310 |  | 178070 |  |  |
  Week 26: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Week 26 |  | 89970 | 503950 |  |  | 220830 | 25020 | 400 | 96180 |  |  |
  Week 30: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
  Week 30 |  | 35210 | 10910 |  |  | 193130 | 29390 | 400 | 36140 |  |  |

12. Secondary Outcome: A Listing, by Arm, of Drug Resistance Test Results and Plasma HIV RNA Levels Among All Participants Who Seroconvert While on Study
Description: Only the listing of drug resistance test by arm among all participants who seroconvert while on study are presented here. See outcome measure 11 for the listing of plasma HIV RNA levels
Time Frame: From Enrollment to week 30 (end of self-administered dosing)
Population: Below, each seroconverted participants' drug resistance test availability was presented. If the number analyzed equal to 0 then it means the resistance test was not done. When the number analyzed equal to 1 and outcome value is 0 then it means no drug resistance was detected, but if the outcome value is 1 then it means drug resistance was detected.
Measure: Number; unit: viral load
Arm/Group | Cape Town, South Africa, Seroconverted Participant #1 | Cape Town, South Africa, Seroconverted Participant #2 | Cape Town, South Africa, Seroconverted Participant #3 | Cape Town, South Africa, Seroconverted Participant #4 | Cape Town, South Africa, Seroconverted Participant #5 | Cape Town, South Africa, Seroconverted Participant #6 | Cape Town, South Africa, Seroconverted Participant #7 | Cape Town, South Africa, Seroconverted Participant #8 | Bangkok, Thailand, Seroconverted Participant #1 | Bangkok, Thailand, Seroconverted Participant #2 | Harlem, United States, Seroconverted Participant #1 | Harlem, United States, Seroconverted Participant #2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
viral load
  Enrollment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 5: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1
  Week 5 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0 |  | 0
  Week 6: number analyzed (Participants) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1
  Week 6 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0
  Week 10: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
  Week 10 |  |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Week 14: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
  Week 14 |  |  | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Week 18: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
  Week 18 |  |  | 0 | 0 | 0 | 1 | 0 | 0 |  |  |  | 0
  Week 22: number analyzed (Participants) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Week 22 |  |  | 0 | 0 | 0 |  | 0 | 0 |  |  |  |
  Week 26: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Week 26 |  |  | 0 |  |  |  |  | 0 |  |  |  |
  Week 30: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Week 30 |  |  |  |  |  |  |  | 0 |  |  |  |

ADVERSE EVENTS:
Time Frame: From week 6 (randomization week) to week 30 (end of self-administered dosing)
Arm/Group | Daily Dosing, Cape Town | Time-driven Dosing, Cape Town | Event-driven Dosing, Cape Town | Daily Dosing, Bangkok | Time-driven Dosing, Bangkok | Event-driven Dosing, Bangkok | Daily Dosing, Harlem | Time-driven Dosing, Harlem | Event-driven Dosing, Harlem
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/59 | 2/60 | 5/60 | 1/59 | 3/59 | 3/59 | 6/60 | 1/60
Other Adverse Events (participants affected / at risk) | 59/59 | 59/59 | 59/60 | 58/60 | 59/59 | 58/59 | 53/59 | 55/60 | 54/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daily Dosing, Cape Town (N=59) | Time-driven Dosing, Cape Town (N=59) | Event-driven Dosing, Cape Town (N=60) | Daily Dosing, Bangkok (N=60) | Time-driven Dosing, Bangkok (N=59) | Event-driven Dosing, Bangkok (N=59) | Daily Dosing, Harlem (N=59) | Time-driven Dosing, Harlem (N=60) | Event-driven Dosing, Harlem (N=60)
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daily Dosing, Cape Town (N=59) | Time-driven Dosing, Cape Town (N=59) | Event-driven Dosing, Cape Town (N=60) | Daily Dosing, Bangkok (N=60) | Time-driven Dosing, Bangkok (N=59) | Event-driven Dosing, Bangkok (N=59) | Daily Dosing, Harlem (N=59) | Time-driven Dosing, Harlem (N=60) | Event-driven Dosing, Harlem (N=60)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 7 | 0 | 1 | 0 | 4 | 4 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0 | 6 | 4 | 4 | 2 | 4 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 7 | 3 | 3 | 1 | 3 | 3 | 2 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 7 | 4 | 6 | 0 | 0 | 0 | 2 | 0 | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 8 | 6 | 7 | 9 | 6 | 3 | 3 | 3 | 4
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alcoholic hangover (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 4 | 1 | 3 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 3 | 0 | 4 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 3 | 3 | 3 | 6 | 1 | 7 | 5 | 4
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 6 | 5 | 1 | 1 | 4 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 10 | 2 | 4 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 2 | 3 | 3 | 4 | 1 | 2 | 0 | 2 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 7 | 8 | 5 | 0 | 0 | 1 | 0 | 1 | 1
Blood sodium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Chlamydial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coital bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 0 | 1 | 4 | 4 | 8
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 4 | 9 | 7 | 9 | 3 | 6 | 6
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 3
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 9 | 13 | 8 | 12 | 13 | 3 | 12
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 9 | 5 | 11 | 8 | 5 | 7 | 6 | 3 | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Dysuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear infection fungal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ejaculation delayed (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejaculation failure (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Episcleritis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 6 | 3 | 8 | 1 | 6 | 1 | 5 | 7 | 6
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 8 | 1 | 3 | 5 | 4 | 7
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 3 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 6 | 3 | 9 | 0 | 2 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Galactorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 4 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital ulceration (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gingival injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Glucose urine (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 2 | 2 | 5 | 0 | 1 | 1 | 0 | 0 | 0
Gonorrhoea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1 | 3 | 0 | 2 | 1 | 1 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hangover (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 24 | 20 | 22 | 13 | 12 | 17 | 9 | 8 | 14
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 4 | 5 | 0 | 0 | 1 | 2 | 4 | 5
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 3 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 4 | 6 | 3 | 2 | 1 | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Lice infestation (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Loss of libido (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 15 | 19 | 22 | 0 | 0 | 0 | 0 | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 3 | 0 | 1 | 3 | 0 | 2 | 2 | 2 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 3 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 6 | 5 | 3 | 8 | 3 | 2 | 4
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 8 | 7
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 26 | 34 | 27 | 6 | 10 | 2
Nausea (Gastrointestinal disorders) | 11 | 12 | 15 | 9 | 2 | 2 | 7 | 8 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 1 | 1 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 2 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oral papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 3 | 27 | 15 | 22 | 4 | 5 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 3 | 3 | 5 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 6 | 5 | 5 | 1 | 2 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penile discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Penis disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Penis injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 3 | 1 | 5 | 1 | 1 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0 | 1 | 7 | 4 | 3
Post-traumatic headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 3 | 4 | 2 | 2 | 3 | 1
Procedural headache (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 1 | 3 | 4 | 3
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 3 | 6 | 5 | 5 | 8 | 7 | 7 | 4
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 0 | 3 | 1 | 0 | 1 | 0 | 2 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 12 | 10 | 11 | 1 | 1 | 2 | 10 | 8 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 1 | 0 | 0 | 2 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pterygium (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 5 | 7 | 4 | 5 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 3 | 7 | 6 | 2 | 1 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 13 | 4 | 3 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sexually transmitted disease (Infections and infestations) | 7 | 8 | 5 | 0 | 0 | 0 | 0 | 0 | 2
Shigella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 1 | 4 | 4 | 5 | 6 | 3 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syphilis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Tinea faciei (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Tinea versicolour (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 3 | 2 | 0 | 1 | 2 | 3 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 1 | 2
Trench foot (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 10 | 0 | 0 | 0 | 0 | 1 | 0
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urethritis chlamydial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urethritis gonococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Urethritis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 8 | 4 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Victim of sexual abuse (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 12 | 13 | 16 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 10 | 2 | 3 | 3 | 1 | 1 | 7 | 4 | 1
Vulvovaginal candidiasis (Infections and infestations) | 2 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study abstracts and publications are subject to HPTN Publication and Public Information Policies and Clinical Trial Agreements between NIAID (DAIDS) and company collaborators. The publication or other disclosure can be delayed for up to thirty additional business days for manuscripts and five business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2013-06-10): https://cdn.clinicaltrials.gov/large-docs/51/NCT01327651/Prot_ICF_000.pdf